Date: 03, 27, 2023

## Informed consent

1- I know that the goals of this research are:

Effects of core stability exercises and cognitive tasks compared to general exercises and cognitive tasks on chronic non-specific back pain

- 2- I know that my participation in this research is completely voluntary and I am not forced to participate in this research.
- 3- I know that even after agreeing to participate in the research, I can withdraw from the research whenever I want.
- 4- My cooperation in this research is as follows:
- -At the specified time, I should visit the rehabilitation faculty for the assessment of posture control.
- -I should go to the rehabilitation faculty at a specified time to receive therapeutic exercises.
- 5- The possible benefits of my participation in this study are as follows:
- -Free low back pain treatment
- -Answering the patient's questions by the research team
- 6- Possible damages and complications of participating in this study are as follows:

No harm threatens me.

- 7- I know that the people involved in this research have kept all the information related to me confidential and they are only allowed to publish the general and group results of this research without mentioning my name and details.
- 8- I know that the research ethics committee can access my information to monitor the observance of my rights
- 9- I know I will not be responsible for any research intervention costs.

- 10- I know that if during and after the research any problem, whether physical or mental, occurs to me due to participating in this research, the treatment of its complications and the related compensation will be the responsibility of the administrator.
- 11- This information and informed consent form have been prepared in two copies, and after signing, one copy will be given to me and the other will be given to the executive.